CLINICAL TRIAL: NCT02735954
Title: Colorado Marijuana Users Health Cohort
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Jewish Health (Other)
Collaborators: Colorado Department of Public Health and Environment (Other Government)
Responsible Party: Sponsor
Other Study IDs: HS 2854
Record Dates: First submitted 2016-01-06; First posted 2016-04-13 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2018-10

CONDITIONS: COPD; Insomnia; Cannabis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Initiation and Maintenance Disorders; Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and urine will be collected and retained for study purposes to look at biomarkers and correlated cannabinoid (THC) levels.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Marijuana Users: Individuals who use marijuana
  Interventions: Other: Marijuana
- Combined Marijuana and Tobacco Users: Individuals who use marijuana and also smoke cigarettes
  Interventions: Other: Marijuana
- Non-Marijuana Users: Individuals who do not use marijuana

INTERVENTIONS:
Other: Marijuana — This is an observational study looking at the effects of marijuana on health, including lung health and sleep.
  Groups: Combined Marijuana and Tobacco Users; Marijuana Users

SUMMARY:
In Colorado, marijuana is currently used for both recreational and medicinal purposes.To learn more about the positive and negative long term medical effects of marijuana use. Information obtained during this study may identify new markers that influence the development of lung diseases such as COPD. The Investigators are also interested in learning more about the effects of marijuana use for insomnia and how it may or may not affect sleep.

DETAILED DESCRIPTION:
In Colorado, marijuana is currently used for both recreational and medicinal purposes. The major active drug is tetrahydrocannabinol (THC). The most common route of use is through inhalation of the combustion products of the dried, buds/flowers from the female plant either rolled in paper (joint) or burned through a screen in a dry or water filled pipe (bong). Increasingly THC is consumed.

The side effects of the inhalation of burned leaves are controversial. The purpose of this proposal is to establish a prospective cohort of heavy marijuana users to evaluate positive and negative long term medical effects of marijuana use. As marijuana has also been reported for use to help treat insomnia, a sub-study will focus on how marijuana is used for sleep disorders and disturbances.

This study will enroll individuals that use marijuana to learn more about long-term health effects. The study involves one visit where participants will complete questionnaires, breathing tests, blood and urine collection. There is a sub-study where eligible participants will also complete an at-home sleep monitoring test. Participants will be contacted multiple times a year for long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Colorado-only study
* Age 21-80 years and one of the categories below
* Marijuana use: use of any cannabis (smoked, vaped, edible, etc.) on average more than 3 days per week for at least 1 year
* Combined marijuana use and Tobacco use (current or former): ≥ 30 pack year cigarette smoking history
* Non-marijuana users

Sleep sub-study:

Enrollment in the main cohort building study and a qualifying score on the Insomnia Severity Index questionnaire

Exclusion Criteria:

* Respiratory disorder other than COPD or asthma
* Lung surgery with removal of a lobe or more or lung volume reduction surgery
* Lung cancer or other cancer under active treatment during past 12 months
* ≥ 30 pack year cigarette smoking history for combined marijuana and cigarette users
* Pregnancy
* Use of antibiotics and/or systemic steroids for any lung infection within the last month
* Inability to use albuterol
* Subject enrolled in COPDGene or SPIROMICS

Sleep sub-study:

* Inability to complete home sleep study

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Colorado investigators are recruiting 1,000 marijuana only users, 1,000 marijuana and tobacco users, and up to 250 non-marijuana users. The sleep sub-study will include up to 218 eligible participants.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-09; Primary Completion 2019-05 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Long term medical effects of marijuana use | measured at baseline visit

SECONDARY OUTCOMES:
Quality of sleep | measured at baseline visit
  physiological parameter and questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States